CLINICAL TRIAL: NCT04797975
Title: A Phase 1/2a Multicenter Randomized Double-blind Placebo-controlled Trial of Off-the-shelf Natural Killer Cells (KDS-1000) as Immunotherapy for Adult Patients With Mild to Moderate COVID-19 Symptoms at Risk for Complications
Brief Title: Off-the-shelf NK Cells (KDS-1000) as Immunotherapy for COVID-19
Status: Withdrawn | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: The sponsor decided to withdraw this study
Sponsor: Kiadis Pharma (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: KNK-COV-001
Record Dates: First submitted 2021-03-12; First posted 2021-03-15 (Actual); Last update posted 2021-08-30 (Actual); Status verified 2021-03

CONDITIONS: Covid19
Keywords: Cell Therapy; COVID-19; Natural Killer Cells; NK Cells; Off-the-shelf
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- KDS-1000 (Experimental): NK cells expanded ex vivo using PM21 membrane particles:
  Interventions: Biological: KDS-1000
- Control (Placebo Comparator): 0.9% Normal Saline
  Interventions: Other: Placebo

INTERVENTIONS:
Biological: KDS-1000 — Non-randomized part of study:
  * At the beginning of each dose level (Cohort), 3 patients will receive KDS-1000. These initial patients will be enrolled in a staggered manner to ensure detection of any early safety signals.
  Randomized part of the study (Can start when there are no safety concerns in the non-randomized cohorts):
  * Cohort 1: Low Dose, 2x10E8 cells/dose
  * Cohort 2: High Dose, 1x10E9 cells/dose
  Arms: KDS-1000
Other: Placebo — 0.9% Normal Saline
  Arms: Control

SUMMARY:
It is hypothesized that immunotherapy with off-the-shelf NK cells (KDS-1000) early in the course of COVID-19 disease is safe and may augment innate immunity, thereby limiting disease progression and improving survival.

DETAILED DESCRIPTION:
Several publications have suggested a potential role of NK cells, an essential part of the early innate response system, in the management of viral infections like COVID-19. Clinical data has shown that COVID-19 disease severity is correlated with a reduction in the number of NK cells, exhaustion of NK cells and the lack of certain mature, potent NK cell phenotypes. The power of NK cells to fight various other viral infections, such as caused by CMV, HBV and hepatitis C virus (HCV), influenza virus and human immunodeficiency virus (HIV) have been well described, with a durable change in the NK cell profile towards those more mature and potent phenotypes in recovered patients. In view of the lack of (functional) NK cells in patients with COVID-19, adoptive NK cell therapy with KDS-1000 cells may improve survival and reduce rates of disease progression from SARS-CoV-2 infection. Adoptive transfer of expanded NK cells (KDS-1000) early in the course of disease may augment innate immunity, thereby limiting disease progression and could confer a survival benefit to patients infected with SARS-CoV-2.

ELIGIBILITY:
Inclusion Criteria:

1. Patients are 18-70 years of age;
2. Patients must have at least one of the following risk factors for developing severe COVID-19 disease:

   1. Age 50 to 70 years;
   2. Obesity (body mass index (BMI) of 30 or greater);
   3. Hypertension;
   4. Current smoker;
   5. Diabetes mellitus (Type 1 or type 2);
   6. Stable cardiac disease.
3. Experiencing symptoms of mild to moderate COVID-19 not requiring supplemental oxygen;
4. Having confirmed infection with SARS-CoV-2, defined as detection of SARS-CoV-2 from nasopharyngeal swab or lower respiratory tract specimen;
5. Karnofsky Performance Score ≥70%;
6. Enrolled within the first 4 days of onset of symptoms;
7. Able and willing to comply with the protocol for duration of the study, including 24 hour hospitalization for study drug administration and monitoring, and compliance with follow-up visit schedule;
8. Signed IRB approved informed consent.

Exclusion Criteria:

1. Patient is at high-risk for severe COVID-19 due to co-morbidities defined as:

   1. Underlying lung disease such as emphysema, chronic lung disease, COPD, asthma, chronic bronchiectasis or respiratory failure requiring baseline oxygen (O2) support;
   2. Immunocompromised host status due to cancer, transplant, or other causes of immunodeficiency;
   3. Immunosuppressive therapy, including but not limited to the following:

      * Corticosteroids (except topical corticosteroids);
      * Interleukin (IL)-6 or Tumor necrosis factor alpha (TNFα) blockade;
      * Other immunotherapies.
2. Patient with the following signs of abnormal organ or bone marrow function as defined below:

   * AST(SGOT) and/or ALT(SGPT) > 3 x upper limit of normal (ULN);
   * Serum (total) bilirubin > 1.5 x ULN;
   * Creatinine Clearance ≤ 30 mL/min (by Modification of Diet in Renal Disease (MDRD) formula);
   * Hemoglobin < 9 g/dL;
   * Thrombocytes ≤ 75.000/uL;
   * Absolute neutrophil count (ANC) ≤ 1.500/uL;
   * Prothrombin time (PT) or activated partial thromboplastin (aPTT) time >1.5 × ULN;
3. Patient has been admitted to the (ICU);
4. Patients with QT prolongation, history of "torsades de pointes" or ventricular arrhythmia (if they are scheduled to receive diphenhydramine);
5. Patient with a known history of allergic reactions to any constituent of the product, including a known history of allergic reactions to cellular products or DMSO;
6. Pregnant (positive pregnancy test) or breast-feeding female patients;
7. Women of childbearing potential who are sexually active and men who have sexual contact with a female of childbearing potential: not willing to use reliable methods of contraception (oral contraceptives, intrauterine device, hormone implants, contraceptive injection or abstinence) up to 90 days post injection of study medication;
8. Participation in other COVID-19 studies involving experimental treatments or vaccines for COVID-19. Participation in other observational studies could be allowed if they do not interfere with protocol compliance or blood draws;
9. Patients with a history or current evidence of alcohol or drug abuse or dependence, or recreational use of illicit drugs including use of medical marijuana;
10. Vulnerable populations such as those currently incarcerated or homeless;
11. Any other condition which in the opinion of the investigator makes the patient ineligible for participation in the study.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2020-12 (Estimated); Primary Completion 2021-04 (Estimated); Study Completion 2021-04 (Estimated)

PRIMARY OUTCOMES:
Determine the safety of KDS-1000 given at low and high doses compared to placebo by collecting the rate and severity of adverse events (AE) | 28 Days
  Rate and severity of AE.

SECONDARY OUTCOMES:
Determine the efficacy KDS-1000 given at low and high doses compared to placebo by COVID-19 specific questionnaire. | 90 Days
  Improvement in COVID-19 disease symptoms/progression of disease.
Determine the efficacy KDS-1000 given at low and high doses compared to placebo by measurement of SARS-CoV-2 clearance. | 28 days
  Determined by real time reverse transcription polymerase chain reaction (rRT-PCR).
Determine the safety of KDS-1000 given at low and high doses compared to placebo by collecting the rate and severity of AE. | 90 Days
  Rate and severity of AE.

IPD SHARING:
Plan to Share IPD: No